CLINICAL TRIAL: NCT02313428
Title: Effects of Topical Oxygen for Diabetic Wounds
Brief Title: Topical Oxygen Therapy for Diabetic Wounds
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment unfulfilled due to lack of staffing.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Chandan Sen, Associate Vice President of Research, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1905092117
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Results first posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Diabetic Foot Ulcers; Wound
Keywords: Diabetic Foot Ulcer; Topical Oxygen Therapy; Medicaid Recipients; Standard of Care; Diabetic Wounds
MeSH Terms: conditions — Diabetic Foot; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard of Care with Topical Oxygen Treatment (Experimental): patients who have a chronic wound, will receive their receive standard treatment plus Topical Oxygen Therapy (Topical Oxygen Chamber for Extremities).
  Interventions: Device: Topical Oxygen Chamber for Extremities
- Standard of Care only (No Intervention): patients that have a chronic wound will receive only their standard of care treatment.

INTERVENTIONS:
Device: Topical Oxygen Chamber for Extremities — Surrounds a limb and applies oxygen topically at a pressure slightly greater than atmospheric pressure to aid healing of chronic skin ulcers
  Other Names: Topical Oxygen Device
  Arms: Standard of Care with Topical Oxygen Treatment

SUMMARY:
This is a pilot study which is intended to collect data to calculate an adequate sample size for a larger registered clinical trial. Eleven subjects were enrolled at The Ohio State University; we intend to enroll 29 more subjects at Indiana University. Due to the small sample size this study will primarily be a feasibility study that will attempt to measure and evaluate differences in the relative theoretical costs of the intervention of topical oxygen therapy on this population and subsequently compare outcomes in areas such as overall health improvements and cost effectiveness.

DETAILED DESCRIPTION:
There are a total of 5 study visits including the initial baseline visit were they will be randomized into one of the 2 groups (comparison or treatment). At the baseline visit the following will be collected; history of the patient, physical examination of the patient including:, digital imaging of the diabetic foot ulcer (DFU) or chronic wound that is input into the WoundMatrix™ software, and the patient will be asked to complete a quality of life questionnaire. Patients will be provided with education regarding diabetes, footwear, and wound care. They will also be given a diary to log their treatments. Patients will return for study visits 2-5 on weeks 4, 8, 12, 16. At study visit 2-5 the research staff will collect digital imaging of the ulcer, review medication, collect previous diary and distribute a new one, and note any wound or health complications. At study visits 1 and 5, the patient will be asked to complete the quality of life questionnaire. These visits will be correlated with their regular scheduled visit at the CWC. If their wound heals before the end of the study, they will be asked to return for study visit 5 (week 16). The patient will complete the at home treatments, including the 90 minute treatment, 4 consecutive days a week, 3 day of no treatment). Study personnel will provide supplies, teach, and give support for the TO device. The study personnel will contact the subject weekly to give support for the treatments.

Participation in this study is expected to add no additional risk to the patient. There is a low risk of local irritation of the skin from application of the Topical Oxygen device for those in the Topical Oxygen Therapy group. This issue is anticipated in the protocol, which specifies appropriate treatment modifications and discontinuation of Topical Oxygen, if it does not improve. If this problem occurs, is expected to be self-limited and of minor significance. Oxygen, although not combustible itself, supports combustion of other flammable materials. The use of oxygen in this protocol is essentially equivalent to that supplied by nasal cannula to patients in hospital or at home. To minimize the risk of fire, the investigators will strictly enforce a 'no smoking' and 'no open flame' policy in any room where Topical Oxygen is utilized. Treatment facilities will comply with local fire ordinances and study personnel will be familiar with fire safety protocols of each facility.

Participants may or may not experience directly benefit from participating in this study. The disease state is highly morbid and typically involves prolonged medical care and multiple surgical procedures. Participants may experience improved healing of their wound as a result of their participation in this study, but there is no guarantee of this. Patients enrolled in the study may also benefit from the close follow-up with study staff and compliance with wound treatment. In addition, the information learned from this research study may lead to a better understanding of diabetic wounds and how they heal, which could lead to better treatment options for patients with diabetic wounds in the future. The application of topical oxygen to diabetic wounds has the potential to dramatically impact the effectiveness of wound healing and to therefore improve limb salvage, decrease infection rates and mortality, and generally improve the quality of life of study participants receiving topical oxygen as well as the general population if efficacy is proved.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Able to give informed consent, willing and able to visit the hospital and CWC for regular treatment and follow-up visits.
* Diabetic
* -Chronic wound OR Foot Ulcer:
* Ulcer present by history ≥ 4 weeks at time of enrollment
* Compliant with standard wound care regimen
* IF foot wound, Wagner grade 1 and 2, OR Wagner grade 3
* Ulcer size: 0.6 cm2 to 20 cm2 and has not decreased in size by more than 30% in previous 2 weeks of the enrollment visit
* Adequate circulatory status, as evidenced by any of the following:
* Ankle Brachial Index (ABI) ≥0.7 - ≥ 1.20
* If ABI non-compressible (ABI >1.2), then toe brachial Index (TBI)>0.5
* SPP > 30mmHg
* TcOM > 30mmHg
* At least 4 weeks since revascularization procedure, if one has been performed
* Able to complete Topical Oxygen Therapy 4 day/week for 16 weeks (must be able to remove existing wound dressing and apply TO2 Boot/treatment, and then re-dress wound)

Exclusion Criteria:

* Ulcer in area of radiation treatment.
* Active malignancy at site of ulcer
* Current treatment with wound VAC or weekly compression dressing
* Untreated infection at site of ulcer (i.e. cellulitis or osteomyelitis)
* If acute osteomyelitis has been diagnosed, patient may be enrolled only after the infection has been controlled. Including:

  1. Debridement of infected bone if necessary
  2. Patient has received at least 2 weeks of appropriate antibiotics
* ABI < 0.7 or > 1.2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandan K. Sen, PhD, Principal Investigator — Indiana University
Locations (1):
- IU Health Methodist Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Fischer BH. Topical hyperbaric oxygen treatment of pressure sores and skin ulcers. Lancet. 1969 Aug 23;2(7617):405-9. doi: 10.1016/s0140-6736(69)90113-5. No abstract available. PMID 4184490
- [Background] Gordillo GM, Roy S, Khanna S, Schlanger R, Khandelwal S, Phillips G, Sen CK. Topical oxygen therapy induces vascular endothelial growth factor expression and improves closure of clinically presented chronic wounds. Clin Exp Pharmacol Physiol. 2008 Aug;35(8):957-64. doi: 10.1111/j.1440-1681.2008.04934.x. Epub 2008 Apr 21. PMID 18430064
- [Background] Heng MCY, Pilgrim JP and Beck FWJ. A simplified technique for hyperbaric oxygen administration for leg ulcers. Clin Res 1982, 30:262A.
- [Background] Heng MC, Pilgrim JP, Beck FW. A simplified hyperbaric oxygen technique for leg ulcers. Arch Dermatol. 1984 May;120(5):640-5. PMID 6721526
- [Background] Kalliainen LK, Gordillo GM, Schlanger R, Sen CK. Topical oxygen as an adjunct to wound healing: a clinical case series. Pathophysiology. 2003 Jan;9(2):81-87. doi: 10.1016/s0928-4680(02)00079-2. PMID 14567939
- [Background] Proposed Rule -General and Plastic Surgery Devices; General Provisions and Classification of 54 Devices, 47 Fed. Reg. 2810-2853 (Jan. 19, 1982).
- [Background] Final Rule -General and Plastic Surgery Devices; General Provisions and Classification of 51 Devices, 53 Fed. Reg. 23856, 23869-23870 (June 24, 1988).
- [Background] Food and Drug Administration, HHS. Medical devices; reclassification of the topical oxygen chamber for extremities. Final rule. Fed Regist. 2011 Apr 25;76(79):22805-7. PMID 21516875
- [Background] Heng MC, Harker J, Bardakjian VB, Ayvazian H. Enhanced healing and cost-effectiveness of low-pressure oxygen therapy in healing necrotic wounds: a feasibility study of technology transfer. Ostomy Wound Manage. 2000 Mar;46(3):52-60, 62. PMID 10788918
- [Background] Heng MC, Harker J, Csathy G, Marshall C, Brazier J, Sumampong S, Paterno Gomez E. Angiogenesis in necrotic ulcers treated with hyperbaric oxygen. Ostomy Wound Manage. 2000 Sep;46(9):18-28, 30-2. PMID 11189538
- [Background] Ware, J.E., Snow, K.K., Kolinski, M., Gandeck, B., 1993. SF-36 Health survey manual and interpretation guide. The Health Institute, New England Medical Centre, Boston, MA.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care With Topical Oxygen Treatment | Standard of Care Only
Started | 2 | 2
Completing 16 wk Visit | 1 | 1
Completed | 1 | 1
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care With Topical Oxygen Treatment | Standard of Care Only | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 44 [44 to 44] | 63 [63 to 63] | 53.5 [44 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Wound Closure
Description: Wound healing rates at 16 weeks of Topical Oxygen Therapy or Standard of Care
Time Frame: baseline and 16 weeks
Measure: Mean (Full Range); unit: cm2
Arm/Group | Standard of Care With Topical Oxygen Treatment | Standard of Care Only
Number analyzed (Participants) | 1 | 1
cm2 | 3.3 [3.3 to 3.3] | 0.00 [0.00 to 0.00]

2. Secondary Outcome: Rate of Amputations
Description: Amputations rates 16 weeks of Topical Oxygen Therapy or Standard of Care
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care With Topical Oxygen Treatment | Standard of Care Only
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

3. Secondary Outcome: Complication Rate
Description: Complication rates (infection) at 16 weeks of Topical Oxygen Therapy or Standard of Care
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care With Topical Oxygen Treatment | Standard of Care Only
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

4. Secondary Outcome: Cost of Care
Description: Post-test health expenditures at 16 weeks of Topical Oxygen Therapy or Standard of Care
Time Frame: 16 weeks
Population: no data could be collected on the cost of measure
Arm/Group | Standard of Care With Topical Oxygen Treatment | Standard of Care Only
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Quality of Life for Subjects- SF-36
Description: QoL data at 16 weeks of Topical Oxygen Therapy or Standard of Care. A cumulative score was calculated based on the QoL responses:
  Note that all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved.
Time Frame: 16 weeks
Measure: Number; unit: percent of total response
Arm/Group | Standard of Care With Topical Oxygen Treatment | Standard of Care Only
Number analyzed (Participants) | 1 | 1
percent of total response | 38.9 | 51.5

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: any new infection or worsening of the wound outcomes that is not anticipated.
Arm/Group | Standard of Care With Topical Oxygen Treatment | Standard of Care Only
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT02313428/Prot_SAP_000.pdf